CLINICAL TRIAL: NCT02821845
Title: Eccentric Motor Control Training to Improve Human Spinal Cord Injury: Observation of Hip and Knee Function
Brief Title: Eccentric Motor Control After SCI
Status: Completed | Type: Observational
Sponsor: Ohio State University (Other)
Collaborators: University of Notre Dame (Other)
Responsible Party: Principal Investigator, Michele Basso, Professor, Ohio State University
Other Study IDs: 2014H0386-2
Record Dates: First submitted 2015-07-11; First posted 2016-07-04 (Estimated); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control: Individuals with no spinal cord injury or other neurological deficits.
- Untrained and Trained SCI Hip and Knee: Individuals with spinal cord injury who have been discharged from a locomotor training program at least 6 months prior to enrollment in this study. Untrained individuals will complete 3 baseline measures and then complete eccentric training which will focus on rehabilitation of the hip joint or knee joint.
  Interventions: Behavioral: Untrained and Trained SCI Hip or Knee

INTERVENTIONS:
Behavioral: Untrained and Trained SCI Hip or Knee — Individuals with SCI will perform downhill walking training 3 times a week for 12 wks with a 4 wk follow-up period. This intervention will be delivered by trained therapists. In order to focus on rehabilitation of hip control or knee control, members of this group will be trained at slow to moderate gait speeds,
  Other Names: DH Hip or Knee
  Groups: Untrained and Trained SCI Hip and Knee

SUMMARY:
This project will characterize lower extremity eccentric muscle function among individuals who have undergone locomotor training after spinal cord injury and will evaluate the effect of downhill training at slow to moderate speeds - targeted to rehabilitation eccentric function of the hip and knee.

DETAILED DESCRIPTION:
Lower extremity eccentric motor control is is critically important for locomotor function but is impaired after spinal cord injury (SCI). Even after treadmill training, preliminary evidence indicates that eccentric deficits persist among individuals with SCI. This proposal aims to characterize eccentric motor control of the muscles about the hip and knee during locomotion and evaluate the efficacy of downhill gait training at slow speeds as an intervention to improve eccentric function of the hip joint and knee joint during walking.

ELIGIBILITY:
Individuals with SCI:

Inclusion Criteria:

* medically approved
* discharged from outpatient rehabilitation for 6 months
* incomplete SCI based on ASIA impairment score (AIS C or D) at neurologic level C1-T10
* ability to take some steps overground and on the treadmill
* 18-90 years old.
* ability to speak English. Note: the quality of life measures have not been validated yet in non-English speaking populations.

Exclusion Criteria:

* evidence of lower motor neuron injury in the legs
* use of botox in the past 3 months
* pre-existing or confounding neurologic conditions (i.e. brain injury, stroke, HIV)
* acute deep vein thrombosis
* skin wounds in regions where harness or hands provide support
* pregnancy. Note: Persons who are pregnant will not be enrolled as exercise tolerance is unknown in these women with SCI.
* cognitive conditions that preclude providing informed consent
* ventilator-dependence as study results will be confounded by mobility limitations imposed by equipment
* persistent orthostatic hypotension (drop of BP >30mmHg in treadmill and harness equipment)
* hospitalization for myocardial infarction, cardiac surgery or congestive heart failure exacerbation within 3 months of enrollment in study
* participation in any other concurrent exercise programs.

Note: Use of anti-spasticity and other medications (dose, frequency) will be monitored throughout training and used as a confounding variable in the analyses.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals from the community that are healthy and without musculoskeletal or orthopedic impairments will serve as healthy case-controls. The individuals with chronic spinal cord injury will come from outpatient clinic referrals and former participants in locomotor training rehabilitation programs.
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2015-06; Primary Completion 2019-10 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in time to complete 6 minutes of level walking (i.e., the 6 minute walk test) | baseline, 12 weeks

SECONDARY OUTCOMES:
Change from baseline in time to complete 10 meters of level walking (i.e., the 10 meter walk test) | baseline, 12 weeks
Change from baseline in peak magnitude of frontal hip loading response as measured by the peak magnitude of frontal hip power absorption during the weight acceptance phase of walking | baseline, 12 weeks

OTHER OUTCOMES:
Change from baseline in Neuromuscular Recovery Scale score | baseline, 12 weeks
Change from baseline in balance function as measured by the Berg Balance Scale score | baseline, 12 weeks
Change from Baseline in SCI specific Quality of Life score | baseline, 12 weeks
Change from second baseline in time to complete 6 minutes of level walking (i.e., the 6 minute walk test) | 12 weeks, 16 weeks
Change from second baseline in time to complete 10 meters of level walking (i.e., the 10 meter walk test) | 12 weeks, 16 weeks
Change from second baseline in peak magnitude of frontal hip loading response as measured by the peak magnitude of frontal hip power absorption during the weight acceptance phase of walking | 12 weeks, 16 weeks
Change from second baseline in quadriceps eccentric contraction capacity as measured by difference in maximum voluntary eccentric knee flexion contraction before and after eccentric exercise targeting the contralateral quadriceps | 12 weeks, 16 weeks
Change from second baseline in Neuromuscular Recovery Scale score | 12 weeks, 16 weeks
Change from second baseline in balance function as measured by Berg Balance Scale score | 12 weeks, 16 weeks
Change from second baseline in SCI specific Quality of Life score | 12 weeks, 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: D. Michele M Basso, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States